CLINICAL TRIAL: NCT00356174
Title: A Prospective Cohort Study of Immune Mechanisms, Genetic Factors, and Clinical and Environmental Characteristics Associated With the Occurrence and Clinical Outcome of Food Allergy (CoFAR2)
Brief Title: An Observational Study of Childhood Food Allergy
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Consortium of Food Allergy Research (Other)
Responsible Party: Sponsor
Other Study IDs: DAIT CoFAR2
Record Dates: First submitted 2006-07-21; First posted 2006-07-25 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Food Hypersensitivity; Peanut Hypersensitivity; Egg Hypersensitivity; Milk Hypersensitivity
Keywords: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity; Egg Hypersensitivity; Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal swab (DNA)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Children with food allergy: 340 longitudinally followed children with egg and/or milk allergy without elevated peanut specific Immunoglobulin E (IgE), less than 5 kUA/L
- Full sibling controls for genetic studies: Approximately 250 not age matched full siblings (i.e., non-step siblings, non-half siblings) will be recruited as an additional control group for genetic studies.
- Full sibling controls for mechanistic studies: Approximately 50 not age matched full siblings (i.e., non-step siblings, non-half siblings) will be recruited as an additional control group for mechanistic studies. A subset of this cohort will be without food allergy,

SUMMARY:
The purpose of this study is to observe the natural course of food allergy, including both the development of peanut allergy in infants at high risk for developing this allergy, and the resolution of both egg and cow's milk allergy.

DETAILED DESCRIPTION:
This observational study will investigate the developmental immunology of peanut, egg, and milk allergy in a cohort of milk- or egg-allergic children who are at risk for peanut allergy. This strategy will help to delineate, compare, and contrast biological markers and immunologic changes associated with the development of peanut allergy and loss of egg and milk allergy, while simultaneously evaluating important clinical and environmental influences likely to account for the recent rise in the prevalence of these allergies. The hallmark of food-allergic disease is the production of food-specific Immunoglobulin E (IgE) antibodies that represent an end result of a T helper 2 (Th2) influenced immune response. Currently, there is only a limited understanding of the mechanisms involved in the developmental course of food allergies. To effectively prevent or reverse the progression of food allergy, immune interventions will be needed. Furthermore, it is likely that successful strategies will need to be directed to those persons at identifiable risk (e.g., who have biomarkers associated with development of peanut allergy).

ELIGIBILITY:
Inclusion Criteria for Children with Food Allergy: Participants who meet all of the following criteria are eligible for enrollment as study participants:

* Atopic dermatitis evaluation
* Either

  1. A convincing clinical history of cow's milk (and/or egg) allergy and a positive prick skin test (≥ 3mm larger than the negative control) to cow's milk (and/or egg, if egg allergy history), or
  2. Moderate to severe atopic dermatitis at the time of enrollment (or by a history prior to removal of milk and/or egg from the maternal (if breastfed) or infant diet) and a positive prick skin test to milk or egg, or
  3. Positive oral food challenge, prior to study entry, to either milk or egg with positive skin test
* Written informed consent from parent/guardian
* Willing to submit specimen for central laboratory plasma peanut IgE

Exclusion Criteria for Children with Food Allergy:

* Participants who meet any of these criteria are not eligible for enrollment as study participants:
* Chronic disease (other than asthma, atopic dermatitis, rhinitis) requiring therapy (e.g., heart disease, diabetes)
* Participation in an interventional study*
* Inability to discontinue antihistamines for routine tests
* Children (other than sibling controls) from families with one child already participating in the observational study
* Confirmed or convincing evidence of peanut allergy

Sibling Inclusion Criteria for Mechanistic Studies:

* No history of food allergy (unrestricted diet), asthma, atopic dermatitis, allergic rhinitis (for blood sample)
* Full sibling of child enrolled in study
* Signed informed consent/assent as applicable

Sibling Exclusion Criteria in Mechanistic Studies:

* Not fulfilling inclusion criteria
* History of chronic anemia
* Disease or medication that impair immune responses

Sibling Inclusion Criteria for Genetic Testing:

* Full sibling of child enrolled in study
* Signed informed consent/assent as applicable

Sibling Exclusion Criteria for Genetic Testing:

* Not fulfilling inclusion criteria

Ages: 3 Months to 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with milk or egg allergy who are at risk for peanut allergy
Sampling Method: Non-Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2006-07; Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Peanut allergy after the age of three years | Year 10
  diagnosed by generally accepted, > 95% accurate, clinical criteria such as oral food challenge.

SECONDARY OUTCOMES:
Resolution of milk allergy after the age of three years | Year 10
  determined by well established criteria with > 95% diagnostic accuracy. Additional (interval analysis) endpoints of egg and milk allergy will be explored in younger children because these allergies may resolve earlier. Common clinical allergy evaluations (e.g., prick skin tests and food-specific IgE antibodies to the 3 targeted foods and common environmental allergens) will be performed and incorporated in the diagnoses of food allergy and atopy.
Resolution of egg allergy after the age of three years | Year 10
  determined by well established criteria with > 95% diagnostic accuracy.
Resolution of peanut allergy after the age of three years | Year 10
  determined by well established criteria with > 95% diagnostic accuracy.
Resolution of a positive test to peanut after the age of three years (suspected allergy category) | Year 10
  determined by well established criteria with > 95% diagnostic accuracy.
Development/persistence of milk allergy after the age of three years | Year 10
  determined by well established criteria with > 95% diagnostic accuracy.
Development/persistence of egg allergy | Year 10
  determined by well established criteria with > 95% diagnostic accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sicherer, MD, Principal Investigator — Jaffe Food Allergy Institute, Icahn School of at Mount Sinai; Hugh Sampson, MD, Principal Investigator — Pediatric Allergy and Immunology, Icahn School of at Mount Sinai
Locations (5):
- United States (5):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - National Jewish Health, Denver, Colorado
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina

REFERENCES:
- [Background] Bjorksten B. Genetic and environmental risk factors for the development of food allergy. Curr Opin Allergy Clin Immunol. 2005 Jun;5(3):249-53. doi: 10.1097/01.all.0000168790.82206.17. PMID 15864084
- [Background] Grundy J, Matthews S, Bateman B, Dean T, Arshad SH. Rising prevalence of allergy to peanut in children: Data from 2 sequential cohorts. J Allergy Clin Immunol. 2002 Nov;110(5):784-9. doi: 10.1067/mai.2002.128802. PMID 12417889
- [Background] Lack G, Fox D, Northstone K, Golding J; Avon Longitudinal Study of Parents and Children Study Team. Factors associated with the development of peanut allergy in childhood. N Engl J Med. 2003 Mar 13;348(11):977-85. doi: 10.1056/NEJMoa013536. Epub 2003 Mar 10. PMID 12637607
- [Background] Sicherer SH, Noone SA, Munoz-Furlong A. The impact of childhood food allergy on quality of life. Ann Allergy Asthma Immunol. 2001 Dec;87(6):461-4. doi: 10.1016/S1081-1206(10)62258-2. PMID 11770692
- [Result] Sicherer SH, Wood RA, Vickery BP, Jones SM, Liu AH, Fleischer DM, Dawson P, Mayer L, Burks AW, Grishin A, Stablein D, Sampson HA. The natural history of egg allergy in an observational cohort. J Allergy Clin Immunol. 2014 Feb;133(2):492-9. doi: 10.1016/j.jaci.2013.12.1041. PMID 24636473
- [Result] Brough HA, Liu AH, Sicherer S, Makinson K, Douiri A, Brown SJ, Stephens AC, Irwin McLean WH, Turcanu V, Wood RA, Jones SM, Burks W, Dawson P, Stablein D, Sampson H, Lack G. Atopic dermatitis increases the effect of exposure to peanut antigen in dust on peanut sensitization and likely peanut allergy. J Allergy Clin Immunol. 2015 Jan;135(1):164-70. doi: 10.1016/j.jaci.2014.10.007. Epub 2014 Nov 18. PMID 25457149
- [Result] Wood RA, Sicherer SH, Vickery BP, Jones SM, Liu AH, Fleischer DM, Henning AK, Mayer L, Burks AW, Grishin A, Stablein D, Sampson HA. The natural history of milk allergy in an observational cohort. J Allergy Clin Immunol. 2013 Mar;131(3):805-12. doi: 10.1016/j.jaci.2012.10.060. Epub 2012 Dec 28. PMID 23273958
- [Result] Fleischer DM, Perry TT, Atkins D, Wood RA, Burks AW, Jones SM, Henning AK, Stablein D, Sampson HA, Sicherer SH. Allergic reactions to foods in preschool-aged children in a prospective observational food allergy study. Pediatrics. 2012 Jul;130(1):e25-32. doi: 10.1542/peds.2011-1762. Epub 2012 Jun 25. PMID 22732173
- [Result] Sicherer SH, Wood RA, Stablein D, Lindblad R, Burks AW, Liu AH, Jones SM, Fleischer DM, Leung DY, Sampson HA. Maternal consumption of peanut during pregnancy is associated with peanut sensitization in atopic infants. J Allergy Clin Immunol. 2010 Dec;126(6):1191-7. doi: 10.1016/j.jaci.2010.08.036. Epub 2010 Oct 28. PMID 21035177
- [Result] Sicherer SH, Wood RA, Stablein D, Burks AW, Liu AH, Jones SM, Fleischer DM, Leung DY, Grishin A, Mayer L, Shreffler W, Lindblad R, Sampson HA. Immunologic features of infants with milk or egg allergy enrolled in an observational study (Consortium of Food Allergy Research) of food allergy. J Allergy Clin Immunol. 2010 May;125(5):1077-1083.e8. doi: 10.1016/j.jaci.2010.02.038. PMID 20451041
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Consortium of Food Allergy Research (CoFAR) — http://www.cofargroup.org/